CLINICAL TRIAL: NCT05213546
Title: Clinical Relevance and Prognostic Outcomes of Different Training Intensities for Cardiac Remodeling in Chronic Heart Failure.
Brief Title: Clinical Relevance of Different Training Intensities in Chronic Heart Failure.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Ahmed Ali Abdeen, Assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HF2021
Record Dates: First submitted 2022-01-16; First posted 2022-01-28 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Chronic Heart Failure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High intensity aerobic training group(HIT) (Active Comparator): 15 patients who received High Intensity aerobic Training in the form of bicycle ergometer exercise for the lower limbs three times /week for three months.
  Interventions: Other: Aerobic exercise training
- Moderate intensity aerobic training group(MIT) (Active Comparator): 15 patients who received moderate Intensity aerobic Training in the form of bicycle ergometer exercise for the lower limbs three times /week for three months.
  Interventions: Other: Aerobic exercise training
- Low intensity aerobic training group(LIT) (Active Comparator): 15 patients who received low Intensity aerobic Training in the form of bicycle ergometer exercise for the lower limbs three times /week for three months
  Interventions: Other: Aerobic exercise training

INTERVENTIONS:
Other: Aerobic exercise training — bicycle ergometer exercise training

SUMMARY:
To determine the efficacy of different aerobic exercise training intensities in patients with chronic heart failure.Forty five eligible male patients with chronic heart failure were randomly assigned into three groups( High intensity , moderate intensity and low intensity)groups .

DETAILED DESCRIPTION:
Forty five eligible male patients with chronic heart failure secondary to ischemic heart disease were selected from National Heart Institute heart failure outpatient clinic , their ages ranged from 50-60 years old and their ejection fraction ranged from 30-40% ,they were randomly assigned into three groups :HIT Group: received High Intensity aerobic Training in the form of bicycle ergometer exercise for the lower limbs three times /week for three months.(n=15) MIT Group: received moderate Intensity aerobic Training in the form of bicycle ergometer exercise for the lower limbs three times /week for three months. .(n=15) LIT Group: received low Intensity aerobic Training in the form of bicycle ergometer exercise for the lower limbs three times /week for three months, Before and after intervention, the following measures were obtained: Echocardiograph parameter (EF%, and left ventricular internal dimension ) , prognostic biomarkers (proBNP), and quality of life .

ELIGIBILITY:
Inclusion Criteria:

* Patients with following criteria were included :

  * All patients ages were between 50 - 60 years old
  * Fractional shortening < 25% and ejection fraction < 40%
  * Sinus rhythm.
  * Heart Failure due to ischemic heart disease.
  * New York Heart Association (NYHA) class II-III.
  * Regular medical treatment.

Exclusion Criteria:

* Patients with following criteria were excluded :

  * Chronic heart failure due to other causes
  * History of pulmonary disease (chronic obstructive lung disease, moderate to severe pulmonary hypertension).
  * Recent acute coronary syndrome or revascularization (3 months).
  * Exercise limited by angina or peripheral arterial occlusive disease;
  * Cerebrovascular or musculoskeletal disease preventing exercise testing or training.
  * Poorly controlled or exercise-induced cardiac arrhythmias
  * Logistic problems to attend regular exercise training sessions. Uncontrolled hypertension.

Ages: 50 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-09-12 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Ejection fraction | change from baseline to after 12 weeks
  represents left ventricular function measured by pulsed echocardiography
pro-brain natriuretic peptide (proBNP) | change from baseline to after 12 weeks
  biomarker for heart failure measured by analysis of venous samples drawn

SECONDARY OUTCOMES:
Minnesota Living With Heart Failure Questionnaire (MLWHF): | change from baseline to after 12 weeks
  Questionnaire for measuring quality of life of heart failure patients

CONTACTS AND LOCATIONS:
Overall Officials: Heba Ahmed Abdeen, PhD, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No